CLINICAL TRIAL: NCT06032000
Title: A Dose-escalation, Double-blinded, Randomized, Placebo-controlled Phase 1 Study to Assess the Safety, Reactogenicity, and Immunogenicity of a SARS-CoV-2 Booster Vaccine (LEM-mR203) in Healthy Adults Aged at 19 to 55 Years
Brief Title: Evaluation of Safety and Immunogenicity of a SARS-CoV-2(Severe Acute Respiratory Syndrome Coronavirus 2) Booster Vaccine (LEM-mR203)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lemonex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LEM-mR203-101
Record Dates: First submitted 2023-08-29; First posted 2023-09-11 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: COVID-19 Infection; COVID-19 Vaccine Adverse Reaction
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: LEM-mR203 vs placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LEM-mR203 (Active Comparator): Drug: LEM-mR203
  An intramuscular single injection prepared by mixing mRNA and DegradaBALL before administration
  Interventions: Biological: LEM-mR203
- Placebo (Placebo Comparator): Drug: 0.9% Sodium Chloride Solution
  An intramuscular single injection prepared before administration
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: LEM-mR203 — mRNA vaccine using Lemonex's Drug Delivery System (DDS), DegradaBALL
  Arms: LEM-mR203
Biological: Placebo — 0.9% Sodium Chloride Solution
  Arms: Placebo

SUMMARY:
A dose-escalation, double-blinded, randomized, placebo-controlled phase 1 study to assess the safety, reactogenicity, and immunogenicity of a SARS-CoV-2 Booster Vaccine (LEM-mR203) in healthy adults aged at 19 to 55 years

DETAILED DESCRIPTION:
The LEM-mR203 is a mRNA vaccine candidate using Lemonex's DDS (Drug Delivery System) named DegradaBALL, and is to be evaluated as a booster vaccine for the prevention of COVID-19 (Coronavirus Disease 2019) in healthy volunteers. DegradaBALL is porous silica nanoparticle-based Drug Delivery System and is resistant to heat and light and stable at room temperature. APIs (Active Pharmaceutical Ingredients) can be loaded by simply mixing into DegradaBALL at the point of use before administration unlike lipid nanoparticles (LNPs) that require drug loading through manufacturing at designated facilities. The LEM-mR203 has been developed to deliver Lemonex's mRNA using DegradaBALL to address the limitations of the existing mRNA COVID-19 vaccines using Lipid Nanoparticle (LNP). The development aims to overcome safety concerns associated with the components of LNP as well as challenges like the ultra-cold storage requirements.

This is the First-In-Human study of LEM-mR203 and consists of two dose cohorts, enrolling healthy adults who will receive a single intramuscular injection of LEM-mR203. The objectives of the trial are to evaluate the safety, reactogenicity, and immunogenicity of LEM-mR203. For each cohort, the first three participants will be dosed with LEM-mR203, followed by a safety review by the DSMB (Data Safety Monitoring Board) before enrolling the remaining participants. The follow-up period will continue for up to 12 months following the administration of a single dose of LEM-mR203.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer aged 19 years or older but less than 55 years at the time of screening.
* Individuals falling into one of the following categories:

  * Those who have completed their primary vaccination with a domestically approved COVID-19 vaccine and have elapsed more than 90 days but less than 48 weeks since the completion of the primary vaccination.
  * Individuals who have completed their primary vaccination and received 1 or more additional doses; these individuals must have elapsed more than 4 months but less than 48 weeks since their last vaccination
* Individuals who do not exhibit clinically significant respiratory symptoms (e.g., cough, sore throat) and do not have clinically significant active lesions on chest X-ray.
* Individuals who agree to use medically accepted contraceptive methods during the entire study period before clinical trials
* Individuals who agree not to donate blood or receive blood transfusions (including whole blood, plasma components, platelet components, and platelet plasma components) during the study period before clinical trials.
* Individuals who can participate in all study visit schedules and comply with all study procedures.
* Individuals who, after receiving detailed explanations about the clinical trial and fully comprehending it, voluntarily decide to participate, and provide written consent before the screening procedure.

Exclusion Criteria:

* Within 72 hours before administration of the investigational medicinal product, individuals with clinically significant respiratory symptoms (e.g., cough, sore throat), acute febrile illness with body temperature exceeding 38℃, suspicion of other infectious diseases, or individuals with symptoms suspected to be caused by other infectious diseases.
* Individuals who tested positive for SARS-CoV-2 genetic test (RT-PCR) or rapid antigen test during the screening.
* Individuals who have not elapsed 90 days since being diagnosed with COVID-19.
* Individuals with positive results in screening tests for Hepatitis B, Hepatitis C, Syphilis (RPR), or HIV conducted during the screening.
* Individuals with a smoking history within 12 weeks prior to administration of the investigational medicinal product or current smokers (smoking up to 10 cigarettes/month may be allowed based on the investigator's judgment ).
* Individuals with a history of malignant tumors within 5 years before administration of the investigational medicinal product.
* Individuals with a history of generalized urticaria within 5 years before administration of the investigational medicinal product.
* Individuals with clinically significant conditions or medical history (e.g., respiratory diseases such as asthma, chronic obstructive pulmonary disease, active tuberculosis; cardiovascular diseases such as congestive heart failure, myocardial infarction, coronary artery disease, uncontrolled hypertension; gastrointestinal diseases such as chronic liver disease, inflammatory bowel disease; hematological and neoplastic diseases, endocrine diseases such as diabetes, hyperthyroidism; genitourinary diseases such as chronic urinary tract infections, chronic renal failure; musculoskeletal diseases such as muscular dystrophy; neurological and psychiatric diseases such as epilepsy, mood disorders, obsessive-compulsive disorder), not limited to the mentioned examples.
* Individuals with a history of solid organ or bone marrow transplantation.
* Individuals with a history of congenital or acquired immunodeficiency diseases or autoimmune diseases.
* Participants who have received any other vaccines within 4 weeks prior to the investigational medicinal product or who have planned to receive other vaccines within 28 days after the administration of the investigational medicinal product are excluded. However, exception applies to influenza vaccines

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Safety and Reactogenicity Assessment | Baseline, 1week, 4week and 3,6 and12 months post a booster injection
  1. Incidence rate of Acute Immediate Adverse Reactions(IAR) within 30 minutes post administration(sentinel group observed for 2 hours)
  2. Incidence rate of solicited local and systemic Adverse Events (AEs) within 7 days post-administration
  3. Incidence rate of unsolicited AEs within up to 28 days post-administration
  4. Incidence rate of Serious Adverse Events (SAEs), Medically Attended Adverse Events (MAAEs), Adverse Events of Special Interest (AESIs) within up to 366 days post-administration

SECONDARY OUTCOMES:
GMT(geometric mean titer) of Anti-SARS-CoV-2 RBD(receptor-binding domain) IgG | Baseline,1,3,6 and 12 months post a booster injection
  GMT of Anti-SARS-CoV-2 RBD IgG from baseline to 1,3,6 and12 months post a booster injection of LEM-mR203, measured by ECLIA(Electrochemiluminescence Immunoassay)
GMFR(geometric mean fold rise) of Anti-SARS-CoV-2 RBD IgG | Baseline,1,3,6 and 12 months post a booster injection
  GMFR of Anti-SARS-CoV-2 RBD IgG from baseline to 1,3,6 and12 months post a booster injection of LEM-mR203, measured by ECLIA
Proportion of participants achieving seroresponse of Anti-SARS-CoV-2 RBD IgG | Baseline,1,3,6 and 12 months post a booster injection
  Proportion of participants achieving seroresponse(SR defined as at least 2-fold increase fro baseline) of Anti-SARS-CoV-2 RBD IgG from baseline to 1,3,6 and 12 months post a booster injection, measured by ECLIA
GMT(geometric mean titer) of neutralizing antibody to the SARS-CoV-2 (kappa variant) | Baseline,1,3,6 and 12 months post a booster injection
  GMT of neutralizing antibody measured by live virus neutralization assay from baseline to 1, 3, 6 and 12 months post a booster injection
GMFR(geometric mean fold rise) of neutralizing antibody to the SARS-CoV-2 (kappa variant) | Baseline,1,3,6 and 12 months post a booster injection
  GMFR of neutralizing antibody measured by live virus neutralization assay from baseline to 1, 3, 6 and 12 months post a booster injection
Proportion of participants achieving seroresponse of neutralizing antibody to the SARS-CoV-2 (kappa variant) | Baseline,1,3,6 and 12 months post a booster injection
  Proportion of participants achieving seroresponse(SR defined as at least 2-fold increase from baseline) of neutralizing antibody measured by live virus from baseline to 1, 3, 6 and 12 months post a booster injection
Cell-mediated Immunity (CMI) | Baseline and 1 month
  INF(Interferon)-γ(gamma) and IL(Interleukin)-4 confirmed using ELISPOT (Enzyme-Linked ImmunoSpot) assay, from baseline to 1 month post a booster injection

CONTACTS AND LOCATIONS:
Overall Officials: Cheolhee Won, PhD, Study Director — Lemonex; In Jin Jang, MD, PhD, Principal Investigator — Seoul National University Hospital Clinical Trials Center
Locations (1):
- Seoul National University Hospital Clinical Trials Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No